CLINICAL TRIAL: NCT01379586
Title: A Phase 1, Single Centre, Three-part, Randomised, Study to Investigate the Safety, Tolerability and Pharmacokinetic Profile of Single and Multiple Ascending Doses of Oral ONO-4053 and the Effects of Food on This Profile in Healthy Male and Female Subjects
Brief Title: A Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of ONO-4053 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4053POE001; Eudra CT No. 2010-023049-31
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-4053; Healthy adult subjects; First time in humans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E (Experimental): ONO-4053
  Interventions: Drug: ONO-4053
- P (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-4053 — Part A: ONO-4053 doses proposed are 1 mg, 3 mg, 10 mg, 30 mg, 100 mg, 300 mg, 600 mg as a single dose administered by mouth once daily
  Arms: E
Drug: Placebo — Placebo to match ONO-4053 tablets dosed in a similar manner to ONO-4053
  Arms: P

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-4053 across ascending single and multiple doses in healthy adult male and female subjects. The secondary objective of the study is to characterize the pharmacokinetic profile of ONO-4053 in healthy adult male and female subjects.

DETAILED DESCRIPTION:
This is a first-in-human study of ONO-4053 in healthy volunteers. This study consists of three parts. Part A will investigate the safety, tolerability and pharmacokinetics when single ascending doses of ONO-4053 are administered in a double-blind manner. Part B will investigate the pharmacokinetics of ONO-4053 in the fed and fasted state in an open-label manner. Part C will investigate the safety, tolerability and pharmacokinetics when multiple ascending doses of ONO-4053 are administered in a double-blind manner. Doses for Part B and C will be determined after data from Part A are available.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian subjects aged 18-45 years inclusive
* Subjects with a body mass index of 19-30 kg/m2 inclusive and who weigh at least 50 kg and no more than 100 kg at screening.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of any clinically significant disease or disorder.
* Current smokers or those that have smoked or used nicotine products within 6 months of the Screening visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-4053 across ascending single and multiple doses using adverse events, vital signs, 12-lead ECG, continuous ECG monitoring and clinical lab tests. | At protocol-specified timepoints before and after study drug administration up to Day 14

SECONDARY OUTCOMES:
Plasma and urine concentrations of ONO-4053 and derived pharmacokinetic parameters | At protocol-specified timepoints before and after study drug administration up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Leeds Clinical Site, Leeds, West Yorkshire, United Kingdom